CLINICAL TRIAL: NCT03170817
Title: Quantitative Rest/Stress Cardiac Perfusion Digital PET/CT: Comparison Between Noninvasive Imaging and Invasive Coronary Angiography.
Brief Title: Quantitative 13N-Ammonia Cardiac Rest/Stress Digital PET/CT
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Guido A. Davidzon, MD, SM, Clinical Assistant Professor, Stanford University
Other Study IDs: IRB 39331
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- N13-ammonia Cardiac Rest/Stress PET/CT: Patients with coronary artery disease (CAD) undergo a Cardiac Perfusion Rest/Stress Digital PET/CT scan using the radiopharmaceutical N13-ammonia and Regadenoson (Lexiscan) to induce pharmacologic stress.
  Interventions: Diagnostic Test: Cardiac Perfusion Rest/Stress Digital PET/CT; Drug: N-13 ammonia; Drug: Regadenoson

INTERVENTIONS:
Diagnostic Test: Cardiac Perfusion Rest/Stress Digital PET/CT — Patients with coronary artery disease undergo a N-13 ammonia rest/stress PET/CT scan.
  These patients are given:
  1. One 5-10 mCI N13-ammonia (13N-NH3) intravenously and undergo a rest digital PET/CT scan of ~20 minute duration.
  2. A dose of 0.4 mg regadenoson (Lexiscan) intravenously over 10 seconds to increase blood flow to the heart
  3. One 5-10 mCi N13-ammonia (13N-NH3) intravenously and undergo a stress digital PET/CT scan of ~20 minute duration
  Total patient time will take approximately up to 120 minutes.
Drug: N-13 ammonia — 5-10 mCi intravenous injection of N-13 ammonia radiopharmaceutical at rest and at stress
Drug: Regadenoson — 0.4 mg/5mL intravenous injection to induce pharmacologic stress (Astellas Pharma US, Inc.)
  Other Names: Lexiscan

SUMMARY:
Accurate measurements from a non-invasive test like myocardial perfusion positron emission tomography/ computed tomography (PET/CT) may decrease the need for invasive procedures such as cardiac catheterization.The investigators wish to see if the measurements from cardiac catheterization can be predicted using a non-invasive 13N-NH3 digital PET/CT scan.

DETAILED DESCRIPTION:
Cardiac imaging using standard-of-care Nuclear Medicine techniques assess the relative radiopharmaceutical distribution from coronary arteries to cardiac tissue. This standard interpretation however, lacks the clinical utility of modern quantitative techniques that are now routinely obtained during cardiac catheterization, such as fractional flow reserve (FFR). Cardiologists routinely base critical management decisions, including the choice for revascularization, stenting, or angioplasty, on these measurements.

Non-invasive measurements of MBF (Myocardial Blood Flow), CFR (Coronary Flow Reserve) and RFR (Relative Flow Reserve) using PET/CT have been investigated, but have yet to reach clinicl use. Given the inherent gains in sensitivity and resolution, digital PET/CT, may allow for a more robust and accurate platform to obtain quantitative measurements of MBF, CFR and RFR which may greatly enhance the clinical utility of cardiac PET/CT for management of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the scan
* Patient has known or suspected coronary artery disease
* Patient has had a recent or will be scheduled for a diagnostic coronary angiogram
* Patient provides written informed consent
* Patient is referred for myocardial perfusion scan
* Patient is capable of complying with study procedures
* Patient is able to remain still for duration of imaging procedure (approximately 60 minutes total for both PET/CT)

Exclusion Criteria:

* Patients who are pregnant or breast feeding
* Patients with contraindications to regadenoson

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stanford Cardiologists will be aware of this ongoing prospective study. Potential participants will be referred to the study by Stanford Cardiology once they are identified by a cardiologist as having intermediate or high risk for a cardiovascular event.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
MBF measurement using PET/CT | an estimated average of 2 hours
  Non-invasive measurements of myocardial blood flow (MBF) in milliliter/minute/gram using PET/CT scanner will be compared to invasive cardiac angiography values (current gold standard). MBF values are obtained using image-derived time activity curves from the left ventricular blood and myocardial tissue regions. These values represent radiotracer exchange between the blood and the tissue over time. The rate of radiotracer uptake into the myocardial tissue provides an estimate of MBF. Processing software will then use the time-activity curves to calculate MBF at rest and at stress.
CFR measurement using PET/CT | an estimated average of 2 hours
  Non-invasive measurements of coronary flow reserve (CFR) using digital PET/CT scanner will be compared to the gold standard evaluation from invasive cardiac angiography. Discrepancy between PET measurements and cardiac angiography results will be reported. CFR is the ratio of MBF at peak blood flow to resting MBF.
RFR measurement using PET/CT | an estimated average of 2 hours
  Non-invasive measurements of relative flow reserve (RFR) using digital PET/CT scanner will be compared to the gold standard evaluation from invasive cardiac angiography. Discrepancy between PET measurements and cardiac angiography results will be reported. RFR is the ratio of MBF during stress in an affected region of the left ventricle (LV) to MBF during stress in a normal region of the LV.

SECONDARY OUTCOMES:
NM Physician diagnostic confidence of 13N-NH3 PET/CT | an estimated average of 2 hours
  Nuclear medicine physician diagnostic confidence will be assessed using a 5-point Likert scale. NM Physicians will compare images obtained from the 13N-NH3 PET/CT to images obtained from single photon emission computed tomography/CT (SPECT/CT).
Overall Exam Time | an estimated average of 2 hours
  Overall study time as counted from initial administration of radiopharmaceutical to completion of image acquisition will be measured and compared to SPECT/CT overall exam time.
Effective radiation dose | an estimated average of 2 hours
  Total radiation dose (measured in mSv) from 13N-NH3 PET/CT will be measured and compared to the dose typically given to patients during standard myocardial perfusion imaging SPECT/CT studies.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Davidzon, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
GE Healthcare is the monitoring entity because GE Healthcare is the Study Sponsor. The monitoring visits will be conducted by a GE Clinical Research Associate (CRA).